CLINICAL TRIAL: NCT03348410
Title: Joint Coordination (GESAM) - Collaboration Project to Facilitate the Transition From Sick Leave to Employment
Brief Title: Joint Coordination to Facilitate the Transition From Sick Leave to Employment
Acronym: GESAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GESAM2017
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Long Term Sick Leave; Absent-mindedness
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Motivational interviewing
  Interventions: Behavioral: Motivational interviewing
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: Motivational interviewing — Motivational interviewing with insurance officer
  Arms: Intervention

SUMMARY:
GESAM is a randomized controlled intervention study that addressed women and men on long-term sick leave in Uppsala County. Participants which are on sick leave due to mental illness and/or pain and were expected to reach the time limit within the in health insurance will be offered to participate in an intervention.

Those how give informed consent will be randomly assigned one of the following groups: 1) informing and motivating intervention with insurance officer 2) control group. The main purpose of the study is to facilitate the return to work (preventing a return to the public health insurance) during the project period.

ELIGIBILITY:
Inclusion Criteria:

* On sick leave
* Risk of losing sick leave compensation

Exclusion Criteria:

* Major mental illness (schizophrenia, bipolar disorder type I, severe social dysfunction/personality disorder)
* Cancer disease

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 193 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
Return to work (RTW) | One year
  Return to work measured as time to participation in the labor force

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Anderzén, PHD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala university, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No